CLINICAL TRIAL: NCT05496439
Title: Study of the Prognosis of Patients With Heart Failure With Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, clinical professor, Chongqing Medical University
Other Study IDs: 2022-08
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: visceral fat area

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study of the prognosis of patients with heart failure with preserved ejection fraction

DETAILED DESCRIPTION:
Obesity is an independent risk factor for heart failure with preserved ejection fraction (HFpEF), however, the impact of visceral fat area (VFA) in patients with HFpEF is unclear. According to established process of patients' selection, a total of 172 patients whose mean age was 72 years were included in this study, and the median follow-up duration was 395.5 days(interquartile range: 207.5 to 535.5 days). All patients were divided into two groups based on the best cut-off value of VFA, and the primary outcome of this study was all-cause death in patients with HFpEF. The aim of this study was to clarify whether VFA has prognostic value in patients with HFpEF by Kaplan-Meier analysis and cox analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged >=18years old;
2. Diagnosed with HFpEF.Diagnostic criteria including:

1）left ventricular ejection fraction ≥50%； 2）with the symptoms and/or signs of heart failure； 3）BNP≥35 pg/mL and/or NTproBNP≥125 pg/mL； 4）at least one additional criterion: relevant structural heart disease(LVH and/or LAE) or diastolic dysfunction

Exclusion Criteria:

1. Age <18 years old；
2. LVEF less than 45% at any time;
3. cancer diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with heart failure with preserved ejection fraction
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
death | The median follow-up time of 395.5 days(interquartile range: 207.5 to 535.5 days)
  all-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No